CLINICAL TRIAL: NCT00153777
Title: Randomized Controlled Trial of 6% Cellulose Sulfate Gel and the Effect on Vaginal HIV Transmission
Brief Title: Cellulose Sulfate and HIV Transmission Among Women
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: IDMC recommendation
Sponsor: CONRAD (Other)
Collaborators: United States Agency for International Development (USAID) (U.S. Federal Agency); Bill and Melinda Gates Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: C03-090
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: HIV Infection
Keywords: HIV prevention; Randomized controlled trial; Women; Sexually transmitted infections; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Cellulose Sulfate gel (6%)

SUMMARY:
The purpose of the study is to determine the effect of cellulose sulfate on the transmission of HIV to women via vaginal intercourse. The secondary objectives are the effect on the transmission of gonorrhea and chlamydia via the same route.

The study hypothesis is that there will be no effect.

DETAILED DESCRIPTION:
Despite the availability of an effective HIV prevention method, i.e. the condom, the epidemic continues growing. There is thus an urgent need for additional HIV prevention methods. One of the possibilities is the use of microbicides, i.e. chemical products which may be used in the vagina or rectum with the potential to prevent HIV infection.

Cellulose sulfate is an HIV entry inhibitor with an in vitro effect on N. gonorrhoeae (NG) and C. trachomatis (CT) and other sexually transmitted organisms.

The study assess its effect on the vaginal transmission of HIV, NG and CT among women at high risk of heterosexual STI infection (defined as having had more than two partners in the last three months and an average of three sexual acts per week).

The study is randomized, triple-blinded, placebo controlled.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old
* an average of at least three vaginal sex acts per week, at least three different partners in the last three months, expecting to continue this behavior
* HIV negative
* willing and able to comply with the protocol

Exclusion Criteria:

* pregnancy
* allergy to latex or spermicides
* intravenous drug user

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1428 (Actual)
Dates: Start 2005-07; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Combined incidence of HIV-1 and HIV-2 in the study. | 1 year

SECONDARY OUTCOMES:
Time-to-first incidental gonococcal or chlamydial infection. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Lut Van Damme, MD, MSc, PhD, Principal Investigator — CONRAD
Locations (5):
- Projet SIDA3, Cotonou, Benin
- India (2):
  - Karnataka Health Promotion Trust, Bangalore
  - YRG Care, Chennai
- Medical Research Council, Durban, South Africa
- Makarere University - Mulago Hospital, Kampala, Uganda

REFERENCES:
- [Background] Crucitti T, Jespers V, Van Damme L, Van Dyck E, Buve A. Vaginal microbicides can interfere with nucleic acid amplification tests used for the diagnosis of Chlamydia trachomatis and Neisseria gonorrhoeae infection. Diagn Microbiol Infect Dis. 2007 Jan;57(1):97-9. doi: 10.1016/j.diagmicrobio.2006.05.010. Epub 2006 Jul 21. PMID 16860515
- [Background] Schwartz JL, Mauck C, Lai JJ, Creinin MD, Brache V, Ballagh SA, Weiner DH, Hillier SL, Fichorova RN, Callahan M. Fourteen-day safety and acceptability study of 6% cellulose sulfate gel: a randomized double-blind Phase I safety study. Contraception. 2006 Aug;74(2):133-40. doi: 10.1016/j.contraception.2006.02.008. Epub 2006 May 2. PMID 16860051
- [Background] El-Sadr WM, Mayer KH, Maslankowski L, Hoesley C, Justman J, Gai F, Mauck C, Absalon J, Morrow K, Masse B, Soto-Torres L, Kwiecien A. Safety and acceptability of cellulose sulfate as a vaginal microbicide in HIV-infected women. AIDS. 2006 May 12;20(8):1109-16. doi: 10.1097/01.aids.0000226950.72223.5f. PMID 16691061
- [Background] Malonza IM, Mirembe F, Nakabiito C, Odusoga LO, Osinupebi OA, Hazari K, Chitlange S, Ali MM, Callahan M, Van Damme L. Expanded Phase I safety and acceptability study of 6% cellulose sulfate vaginal gel. AIDS. 2005 Dec 2;19(18):2157-63. doi: 10.1097/01.aids.0000194797.59046.8f. PMID 16284466
- [Background] Mauck C, Weiner DH, Ballagh S, Creinin M, Archer DF, Schwartz J, Pymar H, Lai JJ, Callahan M. Single and multiple exposure tolerance study of cellulose sulfate gel: a Phase I safety and colposcopy study. Contraception. 2001 Dec;64(6):383-91. doi: 10.1016/s0010-7824(01)00271-2. PMID 11834238
- [Background] Mauck C, Frezieres R, Walsh T, Robergeau K, Callahan M. Cellulose sulfate: tolerance and acceptability of penile application. Contraception. 2001 Dec;64(6):377-81. doi: 10.1016/s0010-7824(01)00270-0. PMID 11834237
- [Background] Anderson RA, Feathergill KA, Diao XH, Cooper MD, Kirkpatrick R, Herold BC, Doncel GF, Chany CJ, Waller DP, Rencher WF, Zaneveld LJ. Preclinical evaluation of sodium cellulose sulfate (Ushercell) as a contraceptive antimicrobial agent. J Androl. 2002 May-Jun;23(3):426-38. PMID 12002445
- [Derived] Guedou FA, Van Damme L, Deese J, Crucitti T, Becker M, Mirembe F, Solomon S, Alary M. Behavioural and medical predictors of bacterial vaginosis recurrence among female sex workers: longitudinal analysis from a randomized controlled trial. BMC Infect Dis. 2013 May 8;13:208. doi: 10.1186/1471-2334-13-208. PMID 23657072
- [Derived] Crucitti T, Fransen K, Maharaj R, Tenywa T, Massinga Loembe M, Murugavel KG, Mendonca K, Abdellati S, Beelaert G, Van Damme L. Obtaining valid laboratory data in clinical trials conducted in resource diverse settings: lessons learned from a microbicide phase III clinical trial. PLoS One. 2010 Oct 27;5(10):e13592. doi: 10.1371/journal.pone.0013592. PMID 21048963
- [Derived] Van Damme L, Govinden R, Mirembe FM, Guedou F, Solomon S, Becker ML, Pradeep BS, Krishnan AK, Alary M, Pande B, Ramjee G, Deese J, Crucitti T, Taylor D; CS Study Group. Lack of effectiveness of cellulose sulfate gel for the prevention of vaginal HIV transmission. N Engl J Med. 2008 Jul 31;359(5):463-72. doi: 10.1056/NEJMoa0707957. PMID 18669425
- See also: Related Info — http://www.conrad.org